CLINICAL TRIAL: NCT00005873
Title: Phase II Study of RFS 2000 (9-Nitro-Camptothecin, 9-NC) in Patients With Relapsed Metastatic Breast Cancer
Brief Title: Nitrocamptothecin in Treating Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067909; SUPERGEN-RFS2000-17; IUMC-9906-11
Record Dates: First submitted 2000-06-02; First posted 2004-04-13 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity and efficacy of nitrocamptothecin in patients with locally recurrent or metastatic breast cancer. II. Determine the duration of response and time to treatment failure in these patients with this treatment regimen. III. Correlate serum levels of nitrocamptothecin and its lactone metabolite with response and toxicity in these patients. IV. Correlate topoisomerase I and II levels with toxicity and response in these patients.

OUTLINE: Patients receive oral nitrocamptothecin daily on days 1-5. Treatment continues weekly for 8 weeks. Patients achieving complete or partial response or stable disease continue therapy in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-43 patients will be accrued for this study within 8-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally recurrent or metastatic breast cancer not amenable to surgery or radiotherapy Measurable or evaluable disease No prior radiotherapy to only target lesion Disease progression after no more than 2 prior chemotherapy treatments for metastatic disease No active CNS metastasis Prior CNS metastasis allowed with no evidence of active disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Not specified Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count greater than 1,500/mm3 Hemoglobin greater than 9.0 g/dL Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST/ALT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN in case of liver metastases) Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Must be able to have daily fluid intake of at least 3 liters No concurrent active infection No other prior malignancy in past 5 years except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior irinotecan, topotecan, or other camptothecin analogues At least 3 weeks since prior chemotherapy Endocrine therapy: No concurrent corticosteroids to control CNS disease Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy Surgery: At least 4 weeks since prior major surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (1):
- SuperGen, Incorporated, Dublin, California, United States